CLINICAL TRIAL: NCT02870777
Title: Minimal Residual Disease-directed Therapy for Low-risk and Intermediate-risk Acute Myeloid Leukemia.
Brief Title: MRD-directed Therapy for Low-risk and Intermediate-risk AML.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Guangzhou First People's Hospital (Other); Zhujiang Hospital (Other); Peking University People's Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRD directed therapy-AML-2016
Record Dates: First submitted 2016-08-14; First posted 2016-08-17 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2019-03

CONDITIONS: Acute Myeloid Leukemia; Minimal Residual Disease
Keywords: MRD; Acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual

STUDY DESIGN:
Intervention Model Description: MRD-directed therapy
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRD-directed therapy (Experimental)
  Interventions: Combination Product: MRD-directed therapy

INTERVENTIONS:
Combination Product: MRD-directed therapy — The purpose of this study is to establish risk stratification based on cytogenetics at diagnosis and MRD analysis after induction chemotherapy and before consolidation chemotherapy to determine whether a MRD directed therapy for low and intermediate AML patients has positive results in terms of overall survival.

SUMMARY:
Acute myeloid leukemia(AML) patients with favorable and intermediate cytogenetics at diagnosis are generally excluded from first-line allo-SCT. However, these patients may eventually relapse in some cases. Our previous study found that stratification of treatment based on cytogenetics and therapeutic response could benefit low and intermediate AML. To further verify the results, we conducted a prospective multi-center study. The purpose of this study is to establish risk stratification based on cytogenetics and minimal-residual-disease (MRD) analysis to determine whether a MRD-directed therapy for low and intermediate AML patients has positive results in terms of overall survival.

ELIGIBILITY:
Inclusion Criteria:

Low-risk and intermediate-risk AML Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure) Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 743 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
disease-free survival (DFS) | 3 year

SECONDARY OUTCOMES:
leukemia relapse rate | 3 year
disease-free survival (DFS) | 3 year
overall survival (OS) | 3 year

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes